CLINICAL TRIAL: NCT00270686
Title: Clinical and Molecular Manifestations of Heritable Disorders of Connective Tissue
Brief Title: Studies of Heritable Disorders of Connective Tissue
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903330; 03-AG-N330
Record Dates: First submitted 2005-12-27; First posted 2005-12-28 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2015-01-02

CONDITIONS: Ehlers-Danlos Syndrome; Stickler Syndrome; Marfan Syndrome
Keywords: Ehlers-Danlos Syndrome; Stickler Syndrome; Marfan Syndrome; Genetics; Aneurysm
MeSH Terms: conditions — Ehlers-Danlos Syndrome; Stickler syndrome, type 1; Marfan Syndrome; Aneurysm

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Heritable disorders of connective tissue are genetic conditions that can affect the skin and other parts of the body. They are related to mutations in genes that are responsible for building tissues. The symptoms differ among disorders. Researchers want to study which genes may be responsible for different disorders. They will be performing a long-term (up to 10 years) study and a study that requires a single visit. These studies will look at how these disorders affect the body and what genes may cause these conditions.

Objectives:

- To perform one-time and long-term studies of people who have heritable disorders of connective tissue.

Eligibility:

- Individuals at least 2 years of age who have or may have a heritable disorder of connective tissue.

Design:

* Participants will be screened with a physical exam, medical history, and blood samples.
* Participants will be on one of two parts of this study. The longitudinal arm will require long-term study over about 10 years. The mutational analysis arm will involve a single visit.
* Longitudinal arm participants must be at least 12 years of age. They will have study visits at regular intervals for up to 10 years. The tests given at these visits may include all or some of the following:
* Blood, saliva, urine, and skin samples
* Heart and lung function tests
* Magnetic resonance imaging scans of the neck, chest, spine, and abdomen
* Other imaging studies such as x-rays, bone density scans, and ultrasounds
* Questionnaires about sleep, pain, and quality of life
* Photographs of affected areas.
* Mutational analysis arm participants will have a single study visit. They will provide blood and saliva samples. They will provide tissue from a skin biopsy. They will also let the researchers take photos of any affected body parts. They will complete questionnaires about sleep, pain, and quality of life.

DETAILED DESCRIPTION:
Heritable disorders of connective tissue are a heterogenous group of genetic conditions caused by defects of extracellular matrix elements such as collagen, elastin, mucopolysaccharides or related biomolecules. The genetic cause of many connective tissue disorders has been elucidated, while others are yet to be discovered or further defined. While clinical diagnostic criteria have been established for several of the connective tissue syndromes, many share features that overlap the known descriptions of other connective tissue disorders. Therefore, further characterization and phenotype/genotype correlation is needed to adequately diagnose and find treatments for these yet-to-be genotyped disorders.

An aim of this work is the examination of the cardiovascular, musculoskeletal and neurological complications of heritable connective tissue disorders (HDCT) and the natural history of these complications. Through mutational analysis for genes known to cause the HDCT, as well as identification of new genes, we will assess the relationship between specific mutations and their associated disease phenotypes. Through the analysis of tissue specimens obtained from patients with HDCT, we will identify the biochemical pathways that lead to connective tissue fragility. We will continue to assess the severity, prevalence, and pattern of pain and related psychological and quality of life dimensions in HDCT.

The resulting understanding of genotype/phenotype correlations and biochemical pathways will enhance our understanding of connective tissue biology. This knowledge has the potential to lead to new treatments for not only patients with HDCT, but also for pathological conditions associated with the weakness of connective tissues in aging.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Individuals and their family members will be offered enrollment if they have an established or suspected diagnosis of Marfan, Stickler, or Ehlers-Danlos syndrome, or Overlap connective tissue disorder.
* Determination of eligibility will be made by review of prior records.
* In some cases, a screening evaluation to establish the diagnosis may be performed subjects may be excluded from further participation if the diagnosis is ruled out. Cytogenetic analysis may be necessary to rule out a chromosomal abnormality that has overlapping features with HDCT.
* Clinical inclusion criteria require: personal or family history of one or more of the following features in a pattern suggestive of a heritable connective tissue disorder: Marfanoid body habitus, aortic dilatation and/or dissection, ectopia lentis, detached retina, vitreous degeneration and/or early onset high myopia, posterior cleft palate, joint laxity and/or dislocation, premature osteoarthritis, skin fragility, striae, easy bruising and/or hyperextensibile skin, pectus excavatum or carinatum, scoliosis, spondylolisthesis and/or dural ectasia, Chiari I Malformation, high frequency sensorineural hearing loss, fibromuscular dysplasia of arteries, aneurysms.

EXCLUSION CRITERIA:

* The only exclusion criterion is inability to provide informed consent, or the absence of a guardian who is authorized to provide informed consent in the case of minor subjects.
* There will be no exclusion based upon age, gender, ethnicity, socioeconomic status, or any other factor except ability to provide informed consent.
* Pregnant and nursing women may be limited in their participation in some aspects of the study (e.g. ionizing radiation exposure or MRI) during the time that they are pregnant or nursing.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 929 (Actual)
Dates: Start 2003-01-21; Study Completion 2015-01-02

PRIMARY OUTCOMES:
Description of natural history of Hereditary Disorders of Connective Tissue (HDCT) | Ongoing
Genetic analysis to identify novel genes that cause HDCT | Ongoing
Biochemical analysis of biospecimens to identify correlations with disease activity and progress | Ongoing
Identification of disease treatment targets | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Nazli B McDonnell, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Background] Ainsworth SR, Aulicino PL. A survey of patients with Ehlers-Danlos syndrome. Clin Orthop Relat Res. 1993 Jan;(286):250-6. PMID 8425354
- [Background] Beighton P, de Paepe A, Danks D, Finidori G, Gedde-Dahl T, Goodman R, Hall JG, Hollister DW, Horton W, McKusick VA, et al. International Nosology of Heritable Disorders of Connective Tissue, Berlin, 1986. Am J Med Genet. 1988 Mar;29(3):581-94. doi: 10.1002/ajmg.1320290316. No abstract available. PMID 3287925
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771